CLINICAL TRIAL: NCT01044706
Title: Randomized, Bioequivalence Study of Bicalutamide 50 mg Tablet and Casodex® 50 mg Tablet Following a 50 mg Dose in Healthy Subjects Under Fed Conditions
Brief Title: Bioequivalence Study of Bicalutamide 50 mg Tablet and Casodex® 50 mg Tablet in Healthy Subjects Under Fed Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kremers Urban Development Company (Industry)
Collaborators: Watson Pharmaceuticals (Industry)
Responsible Party: Benoit Girard, M.D., SFBC Anapharm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 50014
Record Dates: First submitted 2010-01-07; First posted 2010-01-08 (Estimated); Results first posted 2010-03-01 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Healthy
Keywords: Bioequivalency
MeSH Terms: interventions — bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bicalutamide 50 mg Tablet (Experimental): Bicalutamide 50 mg Tablet
  Interventions: Drug: Bicalutamide
- Casodex® 50 mg Tablet (Active Comparator): Casodex® 50 mg Tablet
  Interventions: Drug: Bicalutamide

INTERVENTIONS:
Drug: Bicalutamide — 50 mg Oral Tablet
  Other Names: Casodex®

SUMMARY:
The objective of this study is to compare the rate and extent of absorption of bicalutamide 50 mg tablet (test) versus Casodex® (reference), administered as 1 x 50 mg tablet under fed conditions.

ELIGIBILITY:
Inclusion Criteria:

* Male, non-smoker, 18 years of age and older;
* Capable of consent;
* BMI≥19.0 and <30.0 kg/m2.

Exclusion Criteria:

* Clinically significant illnesses within 4 weeks prior to the administration of the study medication.
* Clinically significant surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which, in the opinion of the Medical Sub-Investigator, would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B, hepatitis C, or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* History of significant alcohol abuse or drug abuse within one year prior to the screening visit.
* Regular use of alcohol within six months prior to the screening visit (more than fourteen units of alcohol per week [1 Unit = 150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol]).
* Use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to heparin, bicalutamide, or other related drugs.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, omeprazole; examples of inhibitors: antidepressants (SSRI), cimetidine, diltiazem, macrolides, imidazoles, neuroleptics, verapamil, fluoroquinolones, antihistamines) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication.
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea, inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological, endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins. garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Use of any tobacco products in the 6 months preceding drug administration.
* Any food allergy, intolerance, restriction or special diet that, in the opinion of the Medical Sub-Investigator, could contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood (excluding the volume of blood that will be drawn during the screening procedures of this study) prior to administration of the study medication as follows:

  * 50 mL to 300 mL of whole blood within 30 days,
  * 301 mL to 500 mL of whole blood within 45 days, or
  * more than 500 mL of whole blood within 56 days prior to drug administration.

Ages: 19 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-05; Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, M.D., Principal Investigator — SFBC Anapharm
Locations (1):
- SFBC Anapharm, Sainte-Foy, Quebec, Canada

RESULTS

PARTICIPANT FLOW:
Recruitment Details: healthy subjects recruited in April 2005 by sfbc Anapharm at 2050, Boul. Rene-Levesque Quest, Saint-Foy, Quebec, Canada G1V 2K8
Pre-assignment Details: This was a single center, bioequivalence, open-label, single-dose, 1-way parallel study
Period: Overall Study
Arm/Group | Bicalutamide 50 mg Tablet | Casodex® 50 mg Tablet
Started | 30 | 30
Completed | 30 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bicalutamide 50 mg Tablet | Casodex® 50 mg Tablet | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 29 | 58
  >=65 years | 1 | 1 | 2
Age Continuous [Mean (Standard Deviation); unit: years] | 40.13 (14.10) | 37.93 (14.41) | 39.03 (14.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 30 | 30 | 60
Region of Enrollment [Number; unit: participants]
  Canada | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: AUC0-144 (Area Under the Concentration-time Curve From Time Zero to 144 Hour Post-dose)
Description: AUC0-144 (area under the concentration-time curve from time zero to 144 hour post-dose)
Time Frame: 144 hour
Population: per protocol
Measure: Geometric Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Bicalutamide 50 mg Tablet | Casodex® 50 mg Tablet
Number analyzed (Participants) | 30 | 30
ng*h/mL | 114386.56 (14285.37) | 105377.55 (11989.86)
Statistical Analysis 1: Comparison: Bicalutamide 50 mg Tablet vs Casodex® 50 mg Tablet; Using GLM procedures in SAS, ANOVA was performed on ln-transformed AUC0-144 at the alpha level of 0.05. Factors incorporated in the model will include: Group, Treatment and Treatment*Group. Intra-subject coefficient of variation (CV%) will be estimated. The ratio of means (T/R) and 90% geometric confidence interval for the ratio of means, based on least-squares means from the ANOVA of the ln-transformed data, will be calculated for AUC0-144 hour; Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference produts. Differences were declared statistically significant at the 5% level (p<0.05); p < 0.05, ANOVA — Differences were declared statistically significant at the 5% level (p<0.05); degrees of freedom 55; ratio of T/R geometric mean x 100 = 108.46, 90% CI 2-sided [102.79 to 114.44], Standard Error of Mean 0.0321 — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean for AUCO-144 and Cmax between the test and reference product fall within the interval of 80-125%

2. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: maximum observed concentration of drug substance in plasma
Time Frame: 144 hour
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bicalutamide 50 mg Tablet | Casodex® 50 mg Tablet
Number analyzed (Participants) | 30 | 30
ng/mL | 1253.60 (138.02) | 1134.86 (122.44)
Statistical Analysis 1: Comparison: Bicalutamide 50 mg Tablet vs Casodex® 50 mg Tablet; Using GLM procedures in SAS, ANOVA was performed on ln-transformed Cmax at the alpha level of 0.05. Factors incorporated in the model will include: Group, Treatment and Treatment*Group. Intra-subject coefficient of variation (CV%) will be estimated. The ratio of means (T/R) and 90% geometric confidence interval for the ratio of means, based on least-squares means from the ANOVA of the ln-transformed data, will be calculated for Cmax; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; p < 0.05, ANOVA — Differences were declared statistically significant at the 5% level (p<0.05); degrees of freedom 56; ratio of T/R geometric mean x 100 = 110.50, 95% CI 2-sided [105.43 to 115.82], Standard Error of Mean 0.0281 — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Arm/Group | Bicalutamide 50 mg Tablet | Casodex® 50 mg Tablet
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 11/30 | 18/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bicalutamide 50 mg Tablet (N=30) | Casodex® 50 mg Tablet (N=30)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pain abdomen (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Pruritus (General disorders) | 1 (1) | 0 (0)
Ecchymosis (Injury, poisoning and procedural complications) | 2 (2) | 2 (2)
Edema inject site (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Hysn inject site (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cramp leg (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain back (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1)
Urine frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This document contains trade secrets and commercial information that is confidential and may not be disclosed to third parties. Persons to whom this study protocol is disclosed must be informed that all the information herein is confidential and may not be further divulged. These restrictions will apply as well to all future communications if deemed privileged or confidential. Publication of the study results may only be allowed with written permission from the Sponsor.